CLINICAL TRIAL: NCT03168061
Title: A Phase 1b/2 Dose-Escalation and Expansion Trial of NC-6300 (Nanoparticle Epirubicin) in Patients With Advanced Solid Tumors or Advanced, Metastatic, or Unresectable Soft Tissue Sarcoma
Brief Title: Dose-Escalation and Expansion Trial of NC-6300 in Patients With Advanced Solid Tumors or Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NanoCarrier Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NC-6300-001
Record Dates: First submitted 2017-04-03; First posted 2017-05-30 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumor; Soft Tissue Sarcoma; Metastatic Sarcoma; Sarcoma
Keywords: advanced solid tumor; unresectable soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — NC 6300

STUDY DESIGN:
Masking Description: open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NC-6300 (Experimental): In Part 1, patients will receive an intravenous infusion of NC-6300 at escalating doses starting at a fixed dose on Day 1 of a 21-day cycle. After enrollment of the initial patient, the first patient in each cohort will not be enrolled until all patients at the immediately lower cohort have completed at least 1 full 21-day cycle. In Part 1, patients will continue to receive treatment until they experience disease progression, experience unacceptable toxicity, or withdraw voluntarily.
  Part 2 will begin after the RPII dose of NC-6300 is identified. All patients in Part 2 will receive NC-6300 at the RPII dose.
  Interventions: Drug: NC 6300

INTERVENTIONS:
Drug: NC 6300 — Part 1: NC-6300 at escalating doses starting at a fixed dose Part 2: NC-6300 at the RPII dose

SUMMARY:
The goal of this study is to find the highest tolerated dose of NC-6300 that can be given to patients with advanced solid tumors or soft tissue sarcoma. The safety and tolerability of the drug will also be studied.

DETAILED DESCRIPTION:
The first part of the study will determine the maximum tolerated dose (MTD), dose-limiting toxicities (DLTs), and the recommended Phase 2 (RPII) dose of NC-6300. The second part of the study will assess the activity and tolerability of NC-6300 in patients with soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* (Part 1 only) Have a histologically/cytologically confirmed diagnosis of advanced solid tumor, including sarcoma that is refractory to standard therapy. (Part 2 only) Have a histologically confirmed diagnosis of advanced, unresectable, or metastatic soft tissue sarcoma not amenable to curative treatment with surgery or radiotherapy.

  * Cohort 1: First-line soft tissue sarcoma of intermediate or high grade. Adjuvant or neoadjuvant chemotherapy allowed if no tumor recurrence for at least 12 months since the last measurement, beginning or end of last chemotherapy.
  * Cohort 2: Soft tissue sarcoma of intermediate or high grade with evidence of disease progression by either CT or MRI scan, or clinical judgment on or after the last cancer therapy within 6 months prior to the start of study treatment. Relapsed or refractory (lack of response) to ≥1 course of systemic therapy regimen(s), excluding adjuvant or neoadjuvant chemotherapy, and is incurable by either surgery or radiation. Patients who have previously received anthracyclines are eligible if cumulative exposure is <375 mg/m2 for doxorubicin and liposomal doxorubicin or <675 mg/m2 for EPI.
* Have measurable disease per RECIST v.1.1.
* Have an ECOG performance status of 0 to 1.
* Have adequate bone marrow reserve defined as:

  * Absolute neutrophil count of at least 1.5 × 109/L,
  * Platelet count of at least 100 × 109/L, and
  * Hemoglobin level of at least 10 g/dL (transfusion is allowed to achieve hemoglobin level of at least 10 g/dL).
* Have adequate liver function defined as:

  * Total serum bilirubin <1.5 × ULN and
  * ALT and AST <2.5 × ULN or, in patients with documented hepatic metastasis, ≤5.0 × ULN.
* Have adequate heart function defined as:

  * LVEF of at least 50%
  * Baseline QTc ≤470 msec and no previous history of QT prolongation while taking other medications.
* Have adequate renal function defined as a creatinine clearance ≥50 mL/minute (calculated according to the formula of Cockcroft and Gault 1976) or serum creatinine <1.5 mg/dL.
* Have reasonably recovered from preceding major surgery as judged by the investigator or have had no major surgery within 4 weeks prior to Day 1 treatment.
* Have stopped previous anticancer therapy for at least 2 weeks or 5 half-lives (whichever is longer) if the immediate prior regimen included only chemotherapy; or 4 weeks or 5 half-lives (whichever is longer) from any therapy with therapeutic biologics and from any type of investigational therapy.
* Women of childbearing potential are will to agree to use 1 of the study defined effective methods of birth control from the time of study entry to 60 days after the final study drug administration
* Women of childbearing potential must have a negative urine pregnancy test at screening, and
* Male patients must use highly effective contraception methods consisting of 2 forms of birth control (at least 1 of which must be a barrier method) starting at screening and continuing throughout the study period and for 60 days after the final study drug administration.

Exclusion Criteria:

* Prior exposure to >375 mg/m2 of doxorubicin or liposomal doxorubicin or ≥675 mg/m2 of EPI.
* Palliative surgery and/or radiation treatment within 30 days prior to date of screening visit.
* (Part 2 only) Current evidence/diagnosis of alveolar soft part sarcoma, extraskeletal myxoid chondrosarcoma, rhabdomyosarcoma, osteosarcoma, gastrointestinal stromal tumor, dermatofibrosarcoma (unless transformed to fibrosarcoma), Ewing's sarcoma, Kaposi's sarcoma, mixed mesodermal tumor, or clear cell sarcomas.
* Evidence of central nervous system metastasis and have not received prior definitive therapy for their lesions.
* Are unable to receive anthracycline therapy due to previous toxicity.
* Have unresolved toxicity from prior radiation, chemotherapy, or other targeted treatment, including investigational treatment, with the exception of alopecia and ≤Grade 1 peripheral neuropathy according to the NCI CTCAE v4.03. Clinical judgment by the investigator is allowed to determine if Grade 1 fatigue at screening is residual toxicity from prior treatment or is a symptom of the patient's general condition or disease. The investigator and Medical Monitor will discuss the eligibility of patients with baseline toxicity.
* Have a history of thrombocytopenia with complications including hemorrhage or bleeding of ≥Grade 2 per NCI CTCAE v4.03 that required medical intervention or have any hemolytic condition or coagulation disorder that would make participation unsafe in the opinion of the investigator.
* Have known hypersensitivity to anthracycline compounds or any excipient in NC-6300.
* Have uncontrolled diabetes or have hypertension requiring more than 3 medications for control of hypertension.
* Have an active, clinically significant serious infection requiring intravenous treatment with antibiotics, antivirals, or antifungals.
* Have signs or symptoms of organ failure, major chronic illnesses other than cancer, or any concomitant medical or social condition that, in the opinion of the investigator, make it undesirable for the patient to participate in the study or that could jeopardize compliance with the protocol.
* Have experienced any of the following within the 6-month period prior to screening: angina pectoris, coronary artery disease or cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%, or severe uncontrolled ventricular arrhythmia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
MTD dose of NC-6300 | up to 7 cycles (21 days/cycle)
RPII dose of NC-6300 | up to 7 cycles (21 days/cycle)

SECONDARY OUTCOMES:
Safety as measured by incidence and severity of TEAEs and laboratory anomalies | through study completion, average 1 year
  To evaluate the overall safety and tolerability of NC-6300 when administered as a single agent
Change in quality of life as measured by EORTC QLQ-C30 | through study completion, average 1 year
  To evaluate the change in health-related quality of life following NC-6300 administration

OTHER OUTCOMES:
Ceoi | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
Cmax | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
Tmax | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
AUC | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
t1/2 | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
Kel | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
CL | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
Vd | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.
Ctrough | through study completion, average 1 year
  To characterize the pharmacokinetics of NC-6300.

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Osada, Study Director — NanoCarrier Co., Ltd.
Locations (7):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California Los Angeles, Santa Monica, California
  - Sarcoma Oncology Research Center, LLC., Santa Monica, California
  - Comprehensive Cancer Centers of Nevada - USOR, Las Vegas, Nevada
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina

REFERENCES:
- [Derived] Riedel RF, Chua V, Moradkhani A, Krkyan N, Ahari A, Osada A, Chawla SP. Results of NC-6300 (Nanoparticle Epirubicin) in an Expansion Cohort of Patients with Angiosarcoma. Oncologist. 2022 Oct 1;27(10):809-e765. doi: 10.1093/oncolo/oyac155. PMID 35920783